CLINICAL TRIAL: NCT06318234
Title: Research Focused on Developing and Assessing a Non-intrusive Diagnostic Approach for Grading Tumor Regression Post-neoadjuvant Treatment in Rectal Cancer, Utilizing 18F-FAPI in Conjunction With FDG PET/MR Imaging.
Brief Title: PET/MR Evaluation of Regression Grading After Neoadjuvant Therapy for Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Xiao Chen (Other)
Responsible Party: Sponsor-Investigator, Xiao Chen, Director of Nuclear Medicine Department, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Other Study IDs: 202435
Record Dates: First submitted 2024-03-05; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Immunotherapy; New assistance; Efficacy evaluation; 18F-FAPI; 18F-FDG; PET/MRI
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — histopathological findings obtained from biopsy or resected surgical specimens
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- After neoadjuvant therapy for rectal cancer: (1) Pathologically confirmed as rectal adenocarcinoma, with baseline clinical staging of T3~4 and/or N+; (2) No distant metastasis; (3) Not receiving chemotherapy or any other anti-tumor treatment before enrollment; (4) Has not received immunotherapy before enrollment and is able to adhere to the protocol during the study period (neoadjuvant therapy of short-term radiotherapy sequential chemotherapy combined with immunotherapy); (5) After neoadjuvant therapy, 18F-FAPI and 18F-FDG PET/MRI imaging were performed within 7 days before surgery, and the two scans were collected over two days; (6) Patient age ≥ 18 years old; (7) The patient voluntarily participates and signs an informed consent form.
  Interventions: Diagnostic Test: 18F-FAPI，18F-FDG

INTERVENTIONS:
Diagnostic Test: 18F-FAPI，18F-FDG — FAPI and FDG combined with PET/MR imaging in patients with rectal cancer after neoadjuvant therapy

SUMMARY:
This project aims to evaluate the role of 18F-FAPI combined with 18F-FDG PET/MRI imaging in quantitatively and accurately evaluating the grading of rectal cancer after SCRT neoadjuvant therapy in patients with advanced rectal cancer as the research object, with postoperative histopathological analysis as the reference index, and to assess the ability of patients to achieve pCR. A diagnostic model and evaluation system will also be constructed.

DETAILED DESCRIPTION:
1. Correlation analysis between the expression levels of FAP and GLUT1 and the degree of tumor regression in rectal cancer

   The study focuses on patients with advanced rectal cancer treated with SCRT neoadjuvant therapy, and conducts immunohistochemical staining of FAP and GLUT1 (glucose transporter 1) on postoperative specimens to evaluate histopathological changes related to the degree of rectal cancer tumor regression. The expression levels of FAP and GLUT1 and the grading of tumor regression are quantitatively analyzed, and their correlation is analyzed to explore the correlation between the expression levels of FAP and GLUT1 in the lesions of neoadjuvant therapy patients and the degree of tumor regression.
2. Construction and validation of a diagnostic model for the degree of tumor regression in rectal cancer after neoadjuvant therapy using 18F-FAPI combined with 18F-FDG PET/MRI imaging

   The patient underwent preoperative 18F-FAPI and 18F-FDG PET/MRI imaging, followed by immunohistochemical staining of FAP and GLUT1 on postoperative specimens and evaluation of histopathological changes related to the degree of rectal cancer tumor regression. The patient's uptake of 18F-FAPI and 18F-FDG (SUVmax, SUVmean, SUVpeak, FAPI metabolic volume, MTV, TBR, TLG), expression levels of FAP and GLUT1, and degree of tumor regression were quantitatively analyzed, and the correlation between the patient's uptake of 18F-FAPI and 18F-FDG and the degree of tumor regression was explored. A graded diagnostic model and evaluation system were constructed to verify their effectiveness.
3. Comparison of the efficacy of PET/MR-TRG and MR-TRG in assessing pTRG after neoadjuvant therapy for rectal cancer

Compare the constructed PET/MR tumor regression grading diagnostic model with the commonly used clinical imaging diagnostic method MRI in evaluating the efficacy, pTRG, and pCR of neoadjuvant therapy for rectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed as rectal adenocarcinoma, with baseline clinical staging of T3~4 and/or N+;
* No distant metastasis;
* Not receiving chemotherapy or any other anti-tumor treatment before enrollment;
* Has not received immunotherapy before enrollment and is able to adhere to the protocol during the study period (neoadjuvant therapy of short-term radiotherapy sequential chemotherapy combined with immunotherapy);
* After neoadjuvant therapy, 18F-FAPI and 18F-FDG PET/MRI imaging were performed within 7 days before surgery, and the two scans were collected over two days;
* Patient age ≥ 18 years old

Exclusion Criteria:

* Pregnant or lactating patients;
* Patients with severe heart disease in clinical practice;
* Organ transplantation requires immunosuppressive therapy and long-term use of hormone therapy;
* Patients with autoimmune diseases;
* Serious uncontrolled recurrent infections or other serious uncontrolled comorbidities;
* The imaging quality is poor and cannot be used for diagnosis and evaluation;
* Fasting blood glucose levels are higher than 11.1 mmol/L;
* Patients with contraindications for MRI examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects the investigators selected are adults who are not restricted by gender.
Sampling Method: Probability Sample
Enrollment: 32 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation efficacy of tumor regression level | Completed within half year after end of the study
  The sensitivity, specificity, positive predictive value (PPV), negative predictive value

SECONDARY OUTCOMES:
expression of FAP | completed within one week after surgery
  Immunohistochemical evaluation of the expression of FAP in postoperative tumor tissue
expression of GLUT1 | completed within one week after surgery
  Immunohistochemical evaluation of the expression of GLUT1 in postoperative tumor tissue
SUV | Completed within one week after PET examination
  Standardized uptake value (SUV) of 18F-FDG and 18F-FAPI for each target lesion of subject or suspected primary tumor or/and metastasis.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Nuclear Medicine, Daping Hospital of Army Medical University, Chongqing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang Y, Shen L, Wan J, Zhang H, Wu R, Wang J, Wang Y, Xu Y, Cai S, Zhang Z, Xia F. Neoadjuvant chemoradiotherapy combined with immunotherapy for locally advanced rectal cancer: A new era for anal preservation. Front Immunol. 2022 Dec 8;13:1067036. doi: 10.3389/fimmu.2022.1067036. eCollection 2022. PMID 36569918